CLINICAL TRIAL: NCT00357955
Title: Combined Behavioral and Pharmacological Intervention for Cardiovascular Risk Reduction in Diabetic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Providence VA Medical Center (U.S. Federal Agency)
Collaborators: Rhode Island Foundation (Other)
Responsible Party: Principal Investigator, Wen-Chih Wu, Staff Cardiologist, Providence VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12733
Record Dates: First submitted 2006-07-24; First posted 2006-07-28 (Estimated); Results first posted 2014-05-13 (Estimated); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Diabetes; Hypertension; Dyslipidemia; Coronary Arteriosclerosis
MeSH Terms: conditions — Diabetes Mellitus; Hypertension; Dyslipidemias; Coronary Artery Disease | interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MEDIC (Experimental): Multidisciplinary education and diabetes intervention for cardiac risk reduction
  Interventions: Behavioral: Behavioral counseling and peer support; Behavioral: Interactive Education; Behavioral: Role modeling; Procedure: Pharmacologic case management
- usual care (No Intervention): usual care

INTERVENTIONS:
Behavioral: Behavioral counseling and peer support — Multidisciplinary education and diabetes intervention for cardiac risk reduction - pharmacist led group intervention
  Arms: MEDIC
Behavioral: Interactive Education — interactive lectures with hands-on learning
  Arms: MEDIC
Behavioral: Role modeling — learning from peers with similar disease and problems
  Arms: MEDIC
Procedure: Pharmacologic case management — provided by clinical pharmacists following pre-established algorithms
  Arms: MEDIC

SUMMARY:
The purpose of this research is to study whether a multidisciplinary education in Diabetes and intervention for cardiac risk reduction in a group setting to modify patient behavior and adjust medications can achieve diabetes guideline goals for glycemia, blood pressure and lipid control.

ELIGIBILITY:
Inclusion Criteria:

* All diabetic veterans with a Hb-A1c between 7.0- 9.0 % within the last 6 months will be eligible for the study

Exclusion Criteria:

* Patients without an Hb-A1c checked within the last 6 months.
* Patients who are unable to attend the group sessions, either because of lack of transportation, psychiatric instability (suicidal, psychotic), or organic brain injury that preclude them from diabetes self-care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2004-08; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Chih Wu, MD, Principal Investigator — Providence VAMC
Locations (1):
- Providence VAMC, Providence, Rhode Island, United States

REFERENCES:
- [Result] Taveira TH, Friedmann PD, Cohen LB, Dooley AG, Khatana SA, Pirraglia PA, Wu WC. Pharmacist-led group medical appointment model in type 2 diabetes. Diabetes Educ. 2010 Jan-Feb;36(1):109-17. doi: 10.1177/0145721709352383. Epub 2009 Dec 4. PMID 19966072
- [Derived] Khatana SA, Taveira TH, Choudhary G, Eaton CB, Wu WC. Change in hemoglobin A(1c) and C-reactive protein levels in patients with diabetes mellitus. J Cardiometab Syndr. 2009 Spring;4(2):76-80. doi: 10.1111/j.1559-4572.2008.00042.x. PMID 19614793

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible patients were identified by a combination of the review of the VA Medical Center's electronic medical record system and referral by primary care providers. Recruitment started July 2004 and enrollment was completed by May 2007.
Pre-assignment Details: Once eligibility confirmed and consent signed, participants were randomized. There were no wash-out or run-in period.
Groups:
- MEDIC: Multidisciplinary education and diabetes intervention for cardiac risk reduction
  Pharmacologic case management : provided by clinical pharmacists following pre-established algorithms
  Behavioral counseling and peer support : Multidisciplinary education and diabetes intervention for cardiac risk reduction - pharmacist led group intervention
  Role modeling : learning from peers with similar disease and problems
  Interactive Education : interactive lectures with hands-on learning
Period: Overall Study
Arm/Group | MEDIC | Usual Care
Started | 64 | 54
Completed | 58 | 51
Not Completed | 6 | 3

BASELINE CHARACTERISTICS:
Population: Age, mean in years; Gender, % male; Baseline level of glycemic control
Groups:
- Total: Total of all reporting groups
Arm/Group | MEDIC | Usual Care | Total
Number analyzed (Participants) | 58 | 51 | 109
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 39 | 20 | 59
  >=65 years | 19 | 31 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (10.3) | 66.8 (10.2) | 64.4 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 0 | 5
  Male | 53 | 51 | 104
Region of Enrollment [Number; unit: participants]
  United States | 58 | 51 | 109

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participans With A1c<7%, LDL Cholesterol <100mg/dL, Systolic Blood Pressure <130mm Hg and Diastolic Blood Pressure <80 mm Hg
Description: The major outcome was the percentage of participants who attain the target goals for A1C, blood pressure,and ldl cholesterol lipids set by the American Diabetes Association guidelines, defined as A1C <7%, SBP <130 mm Hg, diastolic blood pressure (DBP) <80 mm Hg, and LDL cholesterol <100 mg/dL (2.6 mmol/L).
Time Frame: 4 months
Measure: Number; unit: percentage
Groups:
- Usual Care: The standard of care to patients with type 2 diabetes is provided by primary care providers at the VA Medical Center through individual clinic visits. The frequency of these visits for patients with diabetes averages approximately 4 months.usual care
Arm/Group | MEDIC | Usual Care
Number analyzed (Participants) | 58 | 51
percentage
  A1c <7% | 40.4 | 21.6
  Systolic Blood Pressure<130mmHg | 65.5 | 39.9
  Diastolic Blood Pressure<80mmHg | 87.9 | 68.6
  LDL Cholesterol <100mg/dL | 77.2 | 77.5

ADVERSE EVENTS:
Time Frame: Adverse events were documented and reported for the complete study duration of 4 months and 1 month post completion of the study.
Arm/Group | MEDIC | Usual Care
Serious Adverse Events (participants affected / at risk) | 0/58 | 1/51
Other Adverse Events (participants affected / at risk) | 11/58 | 2/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MEDIC (N=58) | Usual Care (N=51)
Hospitalization (Cardiac disorders) | 0 (0) | 1 (1) — was admitted into the hospital for abnormal nonspecific EKG findings from 1/25/06 until 2/1/06
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MEDIC (N=58) | Usual Care (N=51)
Lower Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — seen in the emergency room on 7/25/05 for lower back pain
Syncope (Cardiac disorders) | 1 (1) | 0 (0) — seen in the emergency room and admitted on 7/14/05 for syncope
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) — seen in the emergence room for cough
Cellulitis Abcess (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — was seen in the emergency room on 9/14/05 for cellulitis, hypertension and skin abscess.
Laceration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — was seen in the emergency room on 10/2/05 for a laceration
Blepharitis (Eye disorders) | 1 (1) | 0 (0) — was seen in the emergency room on 8/19/05 for blepheritis
Toe infection (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — was seen in the emergency room on 11/17/05 for a toe infection
Ear ache (Ear and labyrinth disorders) | 1 (1) | 0 (0) — was seen in the emergency room on 1/2/06 for an ear and headache
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — was seen in the emergency room, on 11/19/05 for acute bronchitis
hypertension (Cardiac disorders) | 1 (1) | 0 (0) — was seen in the emergency room on 12/1/05 for hypertension
hematuria (Renal and urinary disorders) | 1 (1) | 0 (0) — was seen in the emergency room on 2/1/06 for hematuria and abdominal pain
rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — was seen in the emergency room on 2/7/06 for rash
hypoglycemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — was seen in the emergency room on 5/29/07 for hypoglycemia

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No